CLINICAL TRIAL: NCT05182333
Title: A Retrospective Study for Congenital Hand and Upper Extremity Malformations in Assiut University Hospital During the Last Twenty Years
Brief Title: Congenital Hand and Upper Extremity Malformations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shady Magdy Makar Salieb, Principle investigator, Assiut University
Other Study IDs: Congenital UL anomalies
Record Dates: First submitted 2021-05-28; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Congenital Limb Anomaly Nos
Keywords: Congenital upper limb anomalies
MeSH Terms: conditions — Limb Deformities, Congenital | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Examination — History taking, examination of upper limb

SUMMARY:
Getting the incidence of upper limb anomalies in our department from 2000 to 2020 and classifying them using IFSSH classification and OMT classification

DETAILED DESCRIPTION:
A retrospective look at the past 20 years illustrated the changes and developments that characterize the world of hand surgery. During these years, old techniques were developed and standardized, new surgical techniques were described, our knowledge improved and illustrated by better classification systems, and new ideas were born that would guide the future of hand surgery. Limb deformities are among the most common birth defects in infants. Over the past 150 years, many classifications of limb abnormalities based on bone morphology and anatomy have been developed.

Congenital anomalies of the hand require consistent and reproducible terminology, and it is a universal language that allows discussion of complex clinical entities, treatment indications and outcome comparisons.

Ideally, the classification of congenital anomalies of the hand will depend on the etiology, giving some indication of the location in the molecular pathway and / or the anatomical location in the developing limb bud where the error occurs and the moment when the fault occurs. The terms should be understandable to geneticists, anatomists, pathologists, and surgeons, and they should allow easy interpretation to parents and, where appropriate, children affected by these conditions. The classification of congenital anomalies of the upper extremity and the important association of these anomalies with systemic disorders and syndromes are described in this study. Depending on the classification, examples are given for each class of anomalies.

ELIGIBILITY:
Inclusion Criteria:

- All patients with congenital upper limb anomalies in last 20 years in Assiut university hospital.

Exclusion Criteria:

* Conditions that were considered to be difficult to correctly classify because of late presentation, a large span of clinical presentation, extremely rare conditions, and conditions difficult to differentiate from traumatic conditions were excluded (ie, congenital radial head dislocation, congenital tumorous conditions, Marfan syndrome)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with congenital upper limb anomalies
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidences of anomalies | Baseline
  Getting the incidences of the upper limb anomalies in upper Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Congenital Hand and Upper Extremity Malformation in Upper Egypt-during the Last Twenty Years

REFERENCES:
- [Background] McCarroll HR. Congenital anomalies: a 25-year overview. J Hand Surg Am. 2000 Nov;25(6):1007-37. doi: 10.1053/jhsu.2000.6457. PMID 11119659
- [Background] Tayel SM, Fawzia MM, Al-Naqeeb NA, Gouda S, Al Awadi SA, Naguib KK. A morpho-etiological description of congenital limb anomalies. Ann Saudi Med. 2005 May-Jun;25(3):219-27. doi: 10.5144/0256-4947.2005.219. PMID 16119523